CLINICAL TRIAL: NCT02734732
Title: Antibiotic Prophylaxis for Transrectal Prostate Biopsy-Ciprofloxacin vs. Trimethoprim/Sulfamethoxazole
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2014---002999---83
Record Dates: First submitted 2016-04-06; First posted 2016-04-12 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Prostate Infection
Keywords: Prostate; Biopsy; Infection; Prophylaxis; Antibiotic
MeSH Terms: conditions — Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination; Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ciprofloxacin (Active Comparator): T. Ciprofloxacin 750mg, single dose immediately prior to prostate biopsy
  Interventions: Drug: Ciprofloxacin
- Trimethoprim/Sulfamethoxazole (Active Comparator): Trimethoprim/Sulfamethoxazole 160mg/800mg immediately prior to prostate biopsy
  Interventions: Drug: Trimethoprim/Sulfamethoxazole

INTERVENTIONS:
Drug: Trimethoprim/Sulfamethoxazole
  Arms: Trimethoprim/Sulfamethoxazole
Drug: Ciprofloxacin
  Arms: Ciprofloxacin

SUMMARY:
This study will examine if a single dose of Ciprofloxacin and Trimethoprim/Sulfamethoxazole are equivalent for prophylaxis immediately prior to prostate biopsy, when a patient has a suspected prostate cancer.

DETAILED DESCRIPTION:
Background: The number of prostate biopsies are estimated to approximately 1.000.000 each year I Europe1. The infection rates after transrectal prostate biopsy are increasing annually2. The most common antibiotic used for prophylaxis is Ciprofloxacin, however, Trimethoprim/Sulfamethoxazole is also a feasible alternative3.

Aim: To evaluate the best antibiotic prophylaxis prior to trans rectal prostate biopsy in low risk patients.

Outcome: Hospitalization for infection within 14 days from biopsy.

Method: By randomization of all eligible patients with low risk of infectious complications. Patient and treating physician is blinded to treatment allocation. By using the nationwide and full coverage national patient register (NPR), mandatory for inpatient care4. All patients can be identified by the Swedish personal identification number5. Both patients related baseline characteristics is gathered through register linkages. To validate the outcome variables, for all patients admitted to hospital within 14 days will be subject for chart review. Comparing all patients from the participating units, having a code specific to trans rectal biopsy, and comparing to the excluded patients as well as included patients, will make a separate exclusion analysis.

The standard operating procedure for randomization is that patients will fill a form and informed consent of participation prior to the planned biopsy. If no exclusion criteria are filled and informed consent obtained, patient will be randomized through a web based randomization program, where only date of biopsy, earlier prostate biopsy, number of biopsies, PSA and prostate size is collected. Other baseline variables will be obtained by cross linkage to the NPR and the National Prostate Cancer Registry. A randomization number is given to all patients at this stage and a key code is established at each participating unit containing every patient randomization number and subsequent personal identification number.

After complete requirement, data will be collected at Västernorrlands Läns Landsting and analyzed according to protocol.

Analysis will be made by logistic regression and point estimates with Single sided 97.5% Confidence Interval. Sample size is calculated to require 2800 patients assuming a 0.5% frequency of infections, able to detect a difference of 0.75% in absolute proportion of infections.

Missing data on outcome variable, received treatment or date of biopsy will be excluded from analysis.

ELIGIBILITY:
Inclusion Criteria:

* Indication for trans rectal prostate biopsy (Physicians discretion)
* Informed consent

Exclusion Criteria:

* Diabetes Mellitus
* Indwelling urinary catheter
* Prior urinary infection (last 6 months)
* Dipstick positive (Nitrites test)
* Allergy to Ciprofloxacin or Trimethoprim/Sulfamethoxazole
* Severe liver disease
* Concomittant use of Tizanidine
* Immunosuppression

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2800 (Estimated)
Dates: Start 2015-04; Primary Completion 2020-04 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Admitted to hospital due to infection | 14 days
  Admission to hospital within 14 days from biopsy

SECONDARY OUTCOMES:
Filled antibiotic prescription | Within 30 days
  A filled prescription within 14 days from biopsy
Positive urinary or blood culture | Within 30 days
  A positive urinary or blood culture obtained within 14 days from biopsy
Any hospital admission | Within 14 days
  Admission to hospital within 14 days from biopsy, regardless of cause
Overall Mortality | Within 90 days
  Overall mortality within 90 days from biopsy
Bacteriological characteristics | Within 30 days
  Resistance patterns and species of bacteria in blood or urinary cultures within 14 days from biopsy
Hospitalisation time | Within 14 days
  Number of days admitted to hospital
Total doses of antibiotics filled | Within 30 days
  The total amount of antibiotics filled
Risk factors for infection | Within 30 days
  Other risk factors for infection apart from exclusion criteria, in baseline variables

CONTACTS AND LOCATIONS:
Overall Officials: Johan Styrke, M.D, Ph.D, Principal Investigator — Umeå University
Locations (5):
- Sweden (5):
  - Östersunds hospital, Östersund, Jämtland County
  - Sundsvalls hospital, Sundsvall, Västernorrland County
  - Ängelholm hospital, Ängelholm
  - Helsingborgs Hospital, Helsingborg
  - Umea University Hospital, Umeå

REFERENCES:
- [Background] Isen K, Kupeli B, Sinik Z, Sozen S, Bozkirli I. Antibiotic prophylaxis for transrectal biopsy of the prostate: a prospective randomized study of the prophylactic use of single dose oral fluoroquinolone versus trimethoprim-sulfamethoxazole. Int Urol Nephrol. 1999;31(4):491-5. doi: 10.1023/a:1007115312039. PMID 10668944
- [Background] Lundstrom KJ, Drevin L, Carlsson S, Garmo H, Loeb S, Stattin P, Bill-Axelson A. Nationwide population based study of infections after transrectal ultrasound guided prostate biopsy. J Urol. 2014 Oct;192(4):1116-22. doi: 10.1016/j.juro.2014.04.098. Epub 2014 May 9. PMID 24813343
- [Background] Wagenlehner FM, Bartoletti R, Cek M, Grabe M, Kahlmeter G, Pickard R, Bjerklund-Johansen TE. Antibiotic stewardship: a call for action by the urologic community. Eur Urol. 2013 Sep;64(3):358-60. doi: 10.1016/j.eururo.2013.05.044. Epub 2013 May 29. PMID 23746854
- [Background] Ludvigsson JF, Andersson E, Ekbom A, Feychting M, Kim JL, Reuterwall C, Heurgren M, Olausson PO. External review and validation of the Swedish national inpatient register. BMC Public Health. 2011 Jun 9;11:450. doi: 10.1186/1471-2458-11-450. PMID 21658213
- [Background] Ludvigsson JF, Otterblad-Olausson P, Pettersson BU, Ekbom A. The Swedish personal identity number: possibilities and pitfalls in healthcare and medical research. Eur J Epidemiol. 2009;24(11):659-67. doi: 10.1007/s10654-009-9350-y. Epub 2009 Jun 6. PMID 19504049